CLINICAL TRIAL: NCT06018805
Title: The Effect of Combined Spinal Epidural Anaesthesia on QTc Interval in Obese and Non-obese Parturients Undergoing Cesarean Section: A Comparative Study
Brief Title: The Effect of Combined Spinal Epidural Anaesthesia on QTc Interval Undergoing Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/408
Record Dates: First submitted 2023-07-24; First posted 2023-08-31 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Mass Index≥30 kg/m2 (Active Comparator): Pregnant women with a Body Mass Index≥30 kg/m2 will be included.
  Interventions: Other: BMI≥30; Combined Spinal Epidural Anesthesia
- Body Mass Index: 18,5 - 24,9 kg/m2 (Active Comparator): Pregnant women with a Body Mass Index between 18.5 and 24.9 kg/m2 will be included.
  Interventions: Other: BMI:18,5-24,9; Combined Spinal Epidural Anesthesia

INTERVENTIONS:
Other: BMI≥30; Combined Spinal Epidural Anesthesia — Combined epidural spinal anesthesia will be performed with the loss of resistance method at constant volume and concentration ( in both patient groups. For QT interval measurements, ECG recordings will be taken before spinal anesthesia, 5 and 30 minutes after the block, and 60 and 120 minutes postoperatively.
  Arms: Body Mass Index≥30 kg/m2
Other: BMI:18,5-24,9; Combined Spinal Epidural Anesthesia — Combined epidural spinal anesthesia will be performed with the loss of resistance method at constant volume and concentration in both patient groups. For QT interval measurements, ECG recordings will be taken before spinal anesthesia, 5 and 30 minutes after the block, and 60 and 120 minutes postoperatively.
  Arms: Body Mass Index: 18,5 - 24,9 kg/m2

SUMMARY:
Cesarean section is the operation to deliver the fetus, placenta and membranes by making an abdominal incision in the uterus. Cesarean section is performed for reasons such as head-pelvis incompatibility, fetal malposition, fetal distress, and previous cesarean section.

The most important side effects of spinal anaesthesia are problems such as hypotension, bradycardia, low back pain, headache, nausea, vomiting, meningitis, meningismus, and urinary retention.

Combined spinal-epidural (BSI) anaesthesia is the application of spinal and epidural anaesthesia together. High-dose local anaesthetics can cause significant hypotension when the epidural block is administered alone. The administration of spinal anaesthesia alone causes changes in arterial resistance, stroke volume, heart rate, cardiac output and arterial blood pressure. Sympathetic blockade leads to arterial vasodilation, and arterial resistance may decrease by 5-20% during spinal anaesthesia.

Due to the increased risk of maternal complications in obese pregnant, fetal morbidity and mortality have increased. In addition, supine hypotension syndrome is a common problem in obese pregnant women. The aim of this study is to compare the change in QTc interval in obese and non-obese term pregnancies planned for elective cesarean section with combined spinal epidural anaesthesia. Thus, it is aimed to develop new protocols that will minimize cardiac pathologies during and after surgery in obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Participants with BMI≥30 and BMI values between 18.5 and 24.9.

Exclusion Criteria:

* allergic to the drugs used in the study,
* who do not accept regional anesthesia,
* body mass index did not meet the inclusion criteria in the study,
* under 150 cm in height,
* who received treatment other than perinatal iron and vitamin drugs,
* smoking or drinking alcohol,
* with a known fetal anomaly,
* with placental disorders such as placenta previa,
* with multiple pregnancy
* have renal or liver disease,
* diagnosed with hypertension or preeclampsia,
* uncooperative and previously treated or currently receiving treatment for a psychiatric disorder
* Mothers who do not want to participate in the study will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
QTc interval | first 2 hour starting from the time of CSE performed.
  The primary aim of this study was to reveal the difference in QTc interval between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Aksoy, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar T, Jha K, Sharan A, Sakshi P, Kumar S, Kumari A. Study of the effect of obesity on QT-interval among adults. J Family Med Prim Care. 2019 May;8(5):1626-1629. doi: 10.4103/jfmpc.jfmpc_168_19. PMID 31198727
- [Background] Song JH, Yang C, Lee W, Kim H, Kim Y, Kim H. QTc interval prolongation due to spinal anesthesia in patients with and without diabetes: an observational study. BMC Anesthesiol. 2022 May 13;22(1):143. doi: 10.1186/s12871-022-01614-8. PMID 35562669